CLINICAL TRIAL: NCT05018481
Title: Mechanism of HA35 in Patients With Alcoholic Liver Disease
Brief Title: HA35 Moderate Alcoholic Hepatitis (AH) Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Srinivasan Dasarathy, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 21-605
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HA35 Placebo Group (Placebo Comparator): 24 study participants will receive the standard of care treatment for AH and a 90-day supply of a placebo to take once a day with breakfast.
  Interventions: Drug: Placebo
- HA35 Treatment Group (Active Comparator): 24 study participants will receive the standard of care treatment for AH and a 90-day supply of a HA35 to take once a day with breakfast.
  Interventions: Drug: Sodium Hyaluronate

INTERVENTIONS:
Drug: Sodium Hyaluronate — Sodium hyaluronate of molecular weight 35kDa will be given in capsule form to study participants
  Other Names: HA35
  Arms: HA35 Treatment Group
Drug: Placebo — A placebo will be given in capsule form to study participants
  Arms: HA35 Placebo Group

SUMMARY:
Eligible participants will be asked to take a placebo/treatment capsule for 90 days and participate in two in-person study visits, one at the start of the 90 days and the second at the completion of study supplement administration. Both visits will include a physical exam, clinical labs, body composition measurements, muscle strength tests, questionnaires, and urine and stool collections. Additionally, a sugar cocktail will be consumed to measure gut permeability and a muscle biopsy will be collected. The day after the visits, you will need to return to drop off the 24-hour urine collection.

Two phone visits will be performed in between the in-person visits at day 30 and 60 where you will be asked a series of questionnaires as well as asked about study supplement compliance.

DETAILED DESCRIPTION:
Written informed consent will be obtained during the baseline visit (day 1). Patients will given a physical exam and a blood test will be obtained if not in their medical chart. The subjects who meet the criteria after the screening visit will have the following procedures: A. Body composition will be quantified by whole-body dual energy X-ray absorptiometry (DEXA), Bioelectric Impedance Analysis (BIA), chair stands, 3 position balance and hand grip strength by dynamometry. B. Muscle biopsy from the lateral portion of vastus lateralis, about 20 cm above knee, C. Questionnaires, D. Blood collection, E. Collection of stool samples, F. Sugar cocktail administration, and G. Urine collection (24 hour)

After baseline measures have been completed, patients will be randomized in a 1:1 ratio to either standard of care (SOC) + HA35 or SOC + placebo (140 mg/d) for a total of 3 months post enrollment.

The subjects will be recalled after 3 months. The visit and the procedures conducted on day 90 will be similar to the baseline study visit.

ELIGIBILITY:
Inclusion Criteria:

• Clinical diagnosis of alcoholic hepatitis defined as:

* Regular consumption of alcohol with an intake of >60 g daily or >420 g weekly on average for men and >40 g daily or >280 g weekly on average for women for 6 months or more

AND

* MELD <21
* Serum total bilirubin >3 mg/dL
* AST >50 IU/I; AST:ALT ratio >1.5; Both AST and ALT <400 IU/I

OR Histologic evidence of AH.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients with gastrointestinal bleeding within 2 weeks
* Active infection (positive blood or ascitic fluid culture)
* Overt encephalopathy
* Renal failure and/or on dialysis
* Medications that alter muscle protein metabolism
* Myopathies
* Other end-stage organ diseases
* Malignancy
* Solid organ or hematopoietic transplantation
* Active alcohol withdrawal or ongoing participation in a Clinical Institute Withdrawal Assessment (CIWA) protocol
* History of recent upper gastrointestinal resection within past 6 months
* Acute or chronic liver disease due to other active causes, in addition to alcoholic liver disease
* Inability to provide consent
* Creatinine >2mg/dL
* Platelets <60,000k/ul
* PT/INR >1.7
* Presence of pedal edema
* Use of anti-platelet/anticoagulation drugs or medications that interfere with blood clotting

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Compare percent change of skeletal muscle mass | Baseline to 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Welch N, Kannan P, Davuluri G, Bellar A, Attaway AH, Mishra S, Cunningham JA, Kumar A, Musich R, Ertugral EG, Agrawal V, Hsu IL, Harford TJ, Weisleder NL, Vachharajani VT, Kothapalli CR, de la Motte CA, Nagy LE, Dasarathy S. Hyaluronan 35 prevents endotoxin-mediated dysregulated skeletal muscle proteostasis during ethanol exposure. Am J Physiol Endocrinol Metab. 2026 Feb 1;330(2):E212-E232. doi: 10.1152/ajpendo.00283.2025. Epub 2026 Jan 6. PMID 41494657